CLINICAL TRIAL: NCT06464978
Title: The Impact of Stapler Reinforcement Patches Compared to Standard Staplers on Postoperative Complications in Gastrojejunostomy: A Multicenter Randomized Controlled Trial
Brief Title: Stapler Reinforcement Patches Compared to Standard Staplers in Gastrojejunostomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanchong Central Hospital (Other Government)
Collaborators: Guang'an Central Hospital (Unknown); Pengan County People's Hospital (Other); Yilong County people's Hospital (Unknown); Nanbu Hospital of County Chinese Medicine (Other); Langzhong People's Hospital (Unknown)
Responsible Party: Principal Investigator, Yunhong Tian, Professor, Nanchong Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20240530
Record Dates: First submitted 2024-06-07; First posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Gastric Cancer; Gastrostomy; Anastomotic Leakage; Postoperative Complications
Keywords: Stapler Reinforcement Patch; Gastrojejunostomy; Randomized Controlled Trial; Surgical Outcomes; Complication Prevention
MeSH Terms: conditions — Stomach Neoplasms; Anastomotic Leak; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the experimental group receiving the stapler reinforcement patches or the control group undergoing standard procedures without reinforcement patches.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcomes assessors will be blinded to the group assignments. Surgeons will be aware of the group assignments but will not disclose this information to the participants or the outcomes assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stapler Reinforcement Patch Group (Experimental): Participants in this group will receive gastrojejunostomy with the use of stapler reinforcement patches.
  Interventions: Device: Stapler Reinforcement Patch
- Standard Stapler Group (Active Comparator): Participants in this group will receive gastrojejunostomy with the use of standard staplers.
  Interventions: Device: Standard Stapler

INTERVENTIONS:
Device: Stapler Reinforcement Patch — Participants in this group will receive gastrojejunostomy with the use of stapler reinforcement patches.
  Arms: Stapler Reinforcement Patch Group
Device: Standard Stapler — Participants in this group will receive gastrojejunostomy with the use of Standard Stapler
  Arms: Standard Stapler Group

SUMMARY:
This is a multi-center, prospective, randomized controlled study aimed at compareing the impact of stapler reinforcement patches versus standard staplers on postoperative complications in gastrojejunostomy.

DETAILED DESCRIPTION:
This study compares stapler reinforcement patches with standard staplers in gastrojejunostomy to reduce postoperative complications. It aims to demonstrate the effectiveness and safety of these patches in preventing anastomotic leakage and other related complications.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 85 years.
* Pathologically diagnosed with gastric cancer and suitable for distal gastrectomy or subtotal gastrectomy.
* ECOG performance status of 0 or 1.
* ASA (American Society of Anesthesiologists) classification of I-III.
* Voluntary signed informed consent from the participant or their legal representative.

Exclusion Criteria:

* Evidence of potential distant metastasis found preoperatively.
* History of other malignancies diagnosed within the past 5 years, or any malignancy treated with chemotherapy or radiotherapy.
* Significant contraindications for surgery (e.g., severe liver or kidney dysfunction).
* Participation in any other clinical trial within the last 6 months.
* Participants or their legal representatives unwilling to sign the informed consent or comply with the study protocol.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Rate of Anastomotic Leakage | 30 days post-surgery
  The incidence of anastomotic leakage within 30 days post-surgery. Anastomotic leakage is defined as the presence of fluid containing enteric content in the abdominal cavity or the appearance of leakage confirmed by imaging or endoscopy.

SECONDARY OUTCOMES:
Rate of Anastomotic Stricture | 3 months post-surgery
  The incidence of anastomotic stricture within 3 months post-surgery. Anastomotic stricture is defined as difficulty in food passage or narrowing confirmed by imaging or endoscopy.
Postoperative Bleeding Rate | 30 days post-surgery
  The incidence of postoperative bleeding within 30 days post-surgery. Postoperative bleeding is defined as the occurrence of bleeding requiring intervention or causing significant hemoglobin drop.
Mortality Rate | 30 days post-surgery
  The rate of mortality within 30 days post-surgery.
Readmission Rate | 3 months post-surgery
  Readmission Rate

CONTACTS AND LOCATIONS:
Locations (1):
- Yunhong Tian, Nanchong, Sichuan, China